CLINICAL TRIAL: NCT05940779
Title: Relationship Between the Risk of Falls and Frailty, and the Effect of a Physical Exercise Program on These Conditions in the Elderly: a Randomized Crossover Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H1504602336419
Record Dates: First submitted 2023-05-31; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-05

CONDITIONS: Frail Elderly Syndrome; Fall

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental)
  Interventions: Other: Therapeutic exercise program
- Control group (No Intervention)

INTERVENTIONS:
Other: Therapeutic exercise program — The intervention is a therapeutic program composed of self-resisted strength exercises, balance training and exercises to improve posture.
  Arms: Exercise group

SUMMARY:
The goal of this randomized crossover clinical trial is to examine the effectiveness of a new therapeutic exercise program in elderly patients with risk of falls and physical fragility. The main questions it aims to answer are:

* If the therapeutic exercise program proposed is a successful treatment for this kind of patients
* If patients at risk of falls also suffer from pre-frailty or frailty, and if they can be treated together with the proposed therapy.

Participants will follow a program consisting of exercises to correct posture, gain strength and contribute to greater balance.

Researchers will compare the therapy and control groups to see if the program increases the percentage of muscle mass of participants, their mobility, balance, quality of life and if they reduce their Fried´s frailty criteria, fear of falling and falls compared to their usual physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling older adults.
* Independent for ambulation.
* With a cognitive state that do not prevent understand the researcher indications.
* Not performing regular physical exercise (only basic activities of daily living, but no other type of intervention).

Exclusion Criteria:

* Contraindication of physical exercise.
* Evident impaired cognitive state.
* Vestibular or central nervous system affection.
* Can´t speak and understand spanish correctly.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | Assessed before the first intervention (baseline).
Timed Up and Go (TUG) | Assessed after the first intervention (3 months later).
Timed Up and Go (TUG) | Assessed after the second intervention (3 months after the previous assessement).
Timed Up and Go (TUG) | Assessed after 3 months from the previous assessement.
Fried frailty criteria | Assessed before the first intervention (baseline).
  The Fried frailty criteria are five: unintentional weight loss, muscular weakness, low resistance or tiredness, slow gait and low level of physical activity.
Fried frailty criteria | Assessed after the first intervention (3 months later).
  The Fried frailty criteria are five: unintentional weight loss, muscular weakness, low resistance or tiredness, slow gait and low level of physical activity.
Fried frailty criteria | Assessed after the second intervention (3 months after the previous assessement).
  The Fried frailty criteria are five: unintentional weight loss, muscular weakness, low resistance or tiredness, slow gait and low level of physical activity.
Fried frailty criteria | Assessed after 3 months from the previous assessement.
  The Fried frailty criteria are five: unintentional weight loss, muscular weakness, low resistance or tiredness, slow gait and low level of physical activity.

SECONDARY OUTCOMES:
Falls and their consequences | Assessed before the first intervention (baseline).
  The number of falls in the last year will be asked.
Falls and their consequences | Every two weeks from date of the first assessement until the date of the study completion, an average of 1 year.
  A follow-up made with phone calls.
Berg Balance Scale (BBS) | Assessed before the first intervention (baseline).
  From 0 to 56. It shows a better balance when the score is higher.
Berg Balance Scale (BBS) | Assessed after the first intervention (3 months later).
  From 0 to 56. It shows a better balance when the score is higher.
Berg Balance Scale (BBS) | Assessed after the second intervention (3 months after the previous assessement).
  From 0 to 56. It shows a better balance when the score is higher.
Berg Balance Scale (BBS) | Assessed after 3 months from the previous assessement.
  From 0 to 56. It shows a better balance when the score is higher.
Falls Efficacy Scale-International (FES-I) | Assessed before the first intervention (baseline).
  From 16 to 64. Higher scores show more concern of falling.
Falls Efficacy Scale-International (FES-I) | Assessed after the first intervention (3 months later).
  From 16 to 64. Higher scores show more concern of falling.
Falls Efficacy Scale-International (FES-I) | Assessed after the second intervention (3 months after the previous assessement).
  From 16 to 64. Higher scores show more concern of falling.
Falls Efficacy Scale-International (FES-I) | Assessed after 3 months from the previous assessement.
  From 16 to 64. Higher scores show more concern of falling.
European Quality of Life-5 Dimensions (EuroQol-5D) | Assessed before the first intervention (baseline).
  It has two parts:
  The first one consists of questions about quality of life with scores from 0 to 1, higher if the quality of life of the patient is higher too.
  The second one is a visual analogic scale (VAS) from 0 (worst quality of life) to 100 (bes quality of life).
European Quality of Life-5 Dimensions (EuroQol-5D) | Assessed after the first intervention (3 months later).
  It has two parts:
  The first one consists of questions about quality of life with scores from 0 to 1, higher if the quality of life of the patient is higher too.
  The second one is a visual analogic scale (VAS) from 0 (worst quality of life) to 100 (bes quality of life).
European Quality of Life-5 Dimensions (EuroQol-5D) | Assessed after the second intervention (3 months after the previous assessement).
  It has two parts:
  The first one consists of questions about quality of life with scores from 0 to 1, higher if the quality of life of the patient is higher too.
  The second one is a visual analogic scale (VAS) from 0 (worst quality of life) to 100 (bes quality of life).
European Quality of Life-5 Dimensions (EuroQol-5D) | Assessed after 3 months from the previous assessement.
  It has two parts:
  The first one consists of questions about quality of life with scores from 0 to 1, higher if the quality of life of the patient is higher too.
  The second one is a visual analogic scale (VAS) from 0 (worst quality of life) to 100 (bes quality of life).
Muscle mass | Assessed before the first intervention (baseline).
  Assessed with and impedance scale.
Muscle mass | Assessed after the first intervention (3 months later).
  Assessed with and impedance scale.
Muscle mass | Assessed after the second intervention (3 months after the previous assessement).
  Assessed with and impedance scale.
Muscle mass | Assessed after 3 months from the previous assessement.
  Assessed with and impedance scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain